CLINICAL TRIAL: NCT06363019
Title: Supporting At-Risk Mothers Across Perinatal Period: A Randomized Controlled Trial
Brief Title: Supporting At-Risk Mothers Across Perinatal Period
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Shefaly Shorey, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/00158
Record Dates: First submitted 2024-03-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Perinatal Depression; Parents; Anxiety; Self Efficacy; Stress; Infant Development
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two-group parallel-armed randomized controlled trial with a pretest and repeated post-test experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers using SMART app (Experimental): The intervention will be delivered via a mobile-based application, the SMART app. The intervention consists of educational material on parenting, pregnancy and managing emotional well-being that mothers are to engage in. Mothers will also participate in the forum with other mother participants. Mothers will also engage in the chat function with a peer volunteer who is an experienced mother. The app is accessible to the mother via the Android or iOS playstore and mother can access anytime in their convenience over 6 months.
  Interventions: Behavioral: Supporting at-risk Mothers Across perinatal period: a Randomized controlled Trial (SMART) mobile application
- Standard Care (No Intervention): This includes routine perinatal visits and check-ups at the hospital or polyclinic the mother is assigned to.

INTERVENTIONS:
Behavioral: Supporting at-risk Mothers Across perinatal period: a Randomized controlled Trial (SMART) mobile application — The intervention is delivered through the SMART mobile application. It contains educational information in audio, visual, article format; on parenting, pregnancy and managing emotional well-being. There is also a peer support feature where participants can speak to experienced mothers via the SMART app. There is also a forum feature where participants can interact with other mothers.
  Arms: Mothers using SMART app

SUMMARY:
The SMART app is a mobile application based psychosocial parenting intervention containing educational materials (articles, videos, audios, podcasts) on parenting, an integrated peer support chat function with experienced mothers and an integrated forum for interaction with other mother participants.

The goal of this interventional study is to test the effectiveness of a mobile-app health based intervention, SMART, mothers in the perinatal period.

The main questions this study aims to answer are:

1. What is the effect of a mobile-based health intervention, SMART, on maternal outcomes?
2. What is the effect of a mobile-based health intervention, SMART, on infant outcomes?
3. What is the cost-effectiveness of using SMART as compared to standard routine care?

Researchers will compare results with a control group that will undergo standard routine care.

DETAILED DESCRIPTION:
This project aims to develop and evaluate a mobile-health application based Supporting at-risk Mothers across perinatal period: A Randomized controlled Trial (SMART) intervention on maternal outcomes such as maternal depression, anxiety and stress, parenting self-efficacy, help-seeking behaviour and attachment and interaction levels , newborn outcomes such as physical, social and emotional development as well as the cost-effectiveness of the intervention.

When compared with those in the control group receiving standard care:

1. mothers receiving SMART intervention will have better: i) emotional well-being (reduced depression, stress, and anxiety); ii) parenting self-efficacy; iii) social support; and iv) attachment, interactions with their newborns and parenting satisfaction.
2. newborns of mothers receiving SMART will have better: i) physical development; ii) social development; and iii) emotional development.
3. It will be more cost-effective to provide SMART than the standard care.

A randomized controlled, two-group pre-test and repeated post-tests, experimental design will be used. Mothers will be randomly assigned to the intervention group, where they will receive the SMART intervention (Access to the mobile App from pregnancy till 6 months postpartum) which includes knowledge-based content with audio and video materials, a peer discussion forum with other mothers, online chat groups with peer volunteer who are experienced mothers plus the standard care. Peer volunteers will be recruited and their role is to provide support to the mother via a weekly chat with the mothers through the SMART application. The control group will receive the standard care provided by the hospitals and polyclinics. The effectiveness of SMART intervention will be measured based on the improvement of maternal depression (primary outcome), stress and anxiety, parenting self-efficacy in newborn care, social support received by mothers, mother-infant attachment, and interactions as well as newborn outcomes including physical, behavioral (social) and emotional development.

Newborn data such as baby gender, order of birth, baby weight and developmental milestones will be collected to examine their development.

ELIGIBILITY:
Inclusion Criteria:

* mothers who (1) are 21 years old to 65 years old; (2) can read and speak English; (3) belong to a vulnerable population due to one or more of the following criteria: i) monthly household income is =/less than SGD 2500 and/or under any low-income support services (referral from social workers) ii) have positive maternal Adverse Childhood Events (ACES) evaluation; iii) single mother; iv) clinically referred by medical professionals or other allied workers for requiring psychosocial support; v) pregnancy or birth of baby diagnosed with congenital malformation/abnormality where baby is 1 year old or less and can be discharged home with mother; vi) mothers with Edinburgh Postnatal Depression Scores (EPDS) =9 (at-risk for depression); and (4) have a smartphone with internet access.

Exclusion Criteria:

* mothers who (1) have chronic physical or mental disorders which would interfere with their ability to participate in the study, and/or (2) gave birth to a baby who needs prolonged hospitalization or NICU support and /or stillborn (3) has a cognitive impairment

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-02-26 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Postnatal depression | Baseline and 6 month, 9month, 12month post childbirth
  Measured via the Edinburgh Postnatal Depression Scale, a 10-item self-reported questionnaire based on a 4-point Likert scale

SECONDARY OUTCOMES:
Infant physical development | 1 month and 6 month at immediate post intervention
  Measured via the Bayley Scale-4th edition
Infant cognitive development | 1 month and 6 month at immediate post intervention
  Measured via the Bayley Scale-4th edition
Infant emotional development | 1 month and 6 month at immediate post intervention
  Measured via the Bayley Scale-4th edition
Anxiety | Baseline and 6 month, 9month, 12month post childbirth
  Measured via the State Trait Anxiety Inventory (STAI), a 40-item self-reported questionnaire based on a 4-point Likert scale
Perceived stress | Baseline and 6 month, 9month, 12month post childbirth
  Measured via the Perceived Stress Scale-10 (PSS-10), a 10-item self-reported questionnaire on a 5 point Likert scale
Perceived social support | Baseline and 6 month, 9month, 12month post childbirth
  Measured via the Perceived Social Support for Parenting (PSSP), a 10-item questionnaire on a 5-point Liker scale
Maternal-infant bonding | 1 month, 6 month, 9 month and 12 month post childbirth
  Measured via the Maternal-Infant Bonding Scale (MIBS), an 8-item self-reported questionnaire on a 4-point Likert scale
Parental satisfaction | Baseline and 6 month, 9month, 12month post childbirth
  Measured via the What Being the Parent of A Baby is Like (WPL), an 11-item self-reported questionnaire on a 9-point Likert scale
Parental efficacy | Baseline and 6 month, 9month, 12month post childbirth
  Measured via a 10-item questionnaire on a 4-point Likert scale
Objective stress | 1 month and 6 month at immediate post intervention
  Measured via salivary cortisol biomarkers obtained through saliva samples
Emotional availability | 1 month and 6 month at immediate post intervention
  Measured through the Emotional Availability Scale (EAS), a 5-dimension framework assessing both the parent and the infant via an observer.
Health services and utilization | Baseline, 1 month, 6 month and 12month post childbirth
  Measured on the Questionnaire on health services and utilization (QHSU)
Infant Physical Development | 1 month, 6 month, 9 month and 12 month post childbirth
  Measured by the Ages and Stages Questionnaire-3
Infant Social Development | 1 month, 6 month, 9 month, 12 month post childbirth
  Measured by the Ages and Stages Questionnaire-3
Infant Social Development | 12 month post childbirth
  Measured by the Brief-Infant and Toddle Social and Emotional Assessment (B-ITSEA)
Infant Social Development | 1 month and 6 month at immediate post intervention
  Measured by the Bayley Scale-4th edition
Infant Emotional Development | 12 month post childbirth
  Measured by the Brief Infant Toddler Social Emotional Assessment (B-ITSEA)

CONTACTS AND LOCATIONS:
Overall Officials: Shefaly Shorey, PhD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - Alice Lee Centre for Nursing Studies, National University of Singapore, Singapore
  - National University of Singapore, Singapore

REFERENCES:
- [Derived] Shah L, Aayisha, Goh YS, Choolani M, Eriksson JG, Chee CYI, Chong SC, Mathews J, Lim LHK, Morelius E, Shorey S. A Window Into Vulnerability and Support: At-Risk Mothers' Perinatal Experiences and Perspectives on mHealth-Based Care. J Adv Nurs. 2025 Oct 18. doi: 10.1111/jan.70292. Online ahead of print. PMID 41109313